CLINICAL TRIAL: NCT05672602
Title: Study of Innovative Biomarkers of Systemic Inflammation in LONG COVID Patients
Brief Title: Biomarkers of LONG COVID (LONG COVID_LCM)
Acronym: LONG COVID_LCM
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Fabio Martelli, Dr, PhD, Molecular Cardiology Laboratory Director, IRCCS Policlinico S. Donato
Other Study IDs: LONG COVID_LCM
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples and peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- LONG COVID patients: Measurement of ncRNAs and cytokines in patients with new diseases or intermittent or permanent symptoms after COVID-19 at the moment of the recruitment
  Interventions: Diagnostic Test: Measurement of ncRNAs and cytokines
- Controls: Measurement of ncRNAs and cytokines in Individuals who have never suffered from COVID-19 at the moment of the recruitment
  Interventions: Diagnostic Test: Measurement of ncRNAs and cytokines
- Asymptomatic LONG COVID patients: Measurement of ncRNAs and cytokines in patients who have never suffered from LONG COVID symptoms or with only resolved symptoms at the moment of the recruitment
  Interventions: Diagnostic Test: Measurement of ncRNAs and cytokines

INTERVENTIONS:
Diagnostic Test: Measurement of ncRNAs and cytokines — Measurement of lncRNAs in PBMCs samples and miRNAs in plasma samples.

SUMMARY:
This observational prospective study is aimed to investigate noncoding RNAs (ncRNAs) such as microRNAs (miRNAs) and long noncoding RNAs (lncRNAs) as potential peripheral blood biomarkers of severity and poor prognosis in COVID-19 patients. Patients with intermittent or permanent symptoms after COVID-19 at the moment of the recruitment were considered affected by LONG COVID disease. In particular, the aim is to clarify if COVID-19 biomarkers remain deregulated similarly in LONG COVID patients. To this purpose, plasma and peripheral blood mononuclear cells (PBMCs) will be collected and patients will be compared to individuals who have never been affected by COVID-19 or asymptomatic LONG COVID patients.

DETAILED DESCRIPTION:
The investigators will collect plasma and PBMCs from consenting subjects. The investigators will evaluate the expression of miRNAs, lncRNAs and cytokines in patients affected by LONG COVID admitted to IRCCS Policlinico San Donato during the acute phase of COVID-19. In particular, miRNAs will be evaluated in plasma samples while lncRNAs in PBMC samples to clarify their potential as biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Previous COVID-19 infection

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to IRCCS Policlinico San Donato during the acute phase of COVID-19
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
LONG COVID biomarkers | Year 1
  Identification of ncRNAs as potential biomarker for the presence of LONG COVID symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No